CLINICAL TRIAL: NCT07018518
Title: Treatment of Pyroptosis-inducible Newcasstle Disease Oncolytic Virus (PIN) Plus Anti-PD1 in Refractory Advanced Primary Hepatocellular Carcinoma---An Open Label Single Arm Phase I Clinical Trial.
Brief Title: PIN in Combination With Anti-PD1 in Previously Treated Primary Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Changping Laboratory (Other)
Responsible Party: Principal Investigator, Han weidong, Director of Biotherapeutic Department, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-096
Record Dates: First submitted 2025-06-05; First posted 2025-06-12 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Hepatocellular Carcinoma; Adult
Keywords: oncolytic viruses; PD-1
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PIN+anti-PD1 (Experimental): 1. Initial treatment phase:
     The combined treatment of PIN and anti-PD1 will be administered for 8 cycles; Unless PD or serious intolerable AEs.
  2. Maintenance treatment phase:
     For patients who completed 8 cycles treatment and obtained effective disease control, if residual tumor lesions are still accessible for local injection, combination therapy will be continued. If no injectable lesion, anti-PD1 will be administrated per 3 weeks till 2 years unless PD or serious intolerable AEs.
  3. Salvage treatment phase:
  For patients who experience disease recurrence or progression 16 weeks after ceasing PIN injection, if there are accessible lesions available for PIN injection, combination therapy will be resumed.
  If specific T cells induced by PIN can be detected in PB when there is no injectable lesion, then the specific T cells are amplified and transfused for salvage therapy.
  Interventions: Biological: PIN +anti-PD1

INTERVENTIONS:
Biological: PIN +anti-PD1 — 1. Initial treatment phase:
     PIN injection frequency:
     day 0 and day 3, per 3 weeks for 8 cycles; PIN injection dosage: Cycle1: 4e9 or 8e9 viral particles of PIN based on the number of injectable lesions, their longest diameter, and the tumor volume capacity .
     Cycle 2~8: 4e9 or 8e9 viral particles of PIN based on the tumor volume's capacity.
     Anti-PD1: day -3, per 3 weeks for 8 cycles;
  2. Maintenance treatment phase:
     No injection lesion: Anti-PD1: day 1, per 3 weeks till 2 years unless PD or serious intolerable AEs.
     Have injection lesion: PIN: 4e9 or 8e9 viral particles based on the tumor volume's capacity, per 6 weeks (within first 24 weeks), then per 8 weeks till 2 years unless unavailability of injection lesion, PD or serious intolerable AEs.
     Anti-PD1: day 1, per 3 weeks till 2 years unless PD or serious intolerable AEs.
  3. Salvage treatment phase: Dosage and frequency of administration refer to the initial treatment phase and maintenance treatment phase.

SUMMARY:
In this single-center,open-label, phase I study, the safety and efficacy of PIN in combination with programmed cell death protein antibody (anti-PD1) therapeutic regimen will be evaluated in patients with refractory primary advanced hepatocellular carcinoma(HCC) . A total of 25 to 30 patients are planned to be enrolled and receive PIN plus anti-PD1 combined treatment. It aims to: 1).assess the safety and antitumor effects of the above combined treatment regimen. 2).detect the dynamic changes and molecular characteristics of PIN-induced CD8+ T cells with special phenotype in peripheral blood (PB) and transformation of tumor microenvironment (TME) after the treatment with PIN. 3).evaluate the immunological or clinical predictive biomarkers for toxicity and efficacy.

DETAILED DESCRIPTION:
Currently, systemic therapy for advanced primary HCC mainly relies on targeted therapy and immunotherapy.However,after disease progression, patients often have limited treatment options and poor prognosis.Therefore, no standard therapies beyond second-line are recommended, highlighting the urgent need for innovative treatments.

Several clinical studies have found that oncolytic viruses (OVs) can provide clinical benefits to patients with various malignant tumors, including advanced HCC.To date, there are hundreds of projects in clinical trial stages, especially in recent years, new generations of OVs developed or in clinical stages have shown better safety and stronger anti-tumor capabilities. Through genetic engineering, OVs can express target genes that have anti-tumor effects, such as granulocyte-macrophage colonystimulating factor (GM-CSF), interleukin-12(IL-12),etc, further enhancing their anti-tumor effects. Despite these advances, how to obtain a more durable antitumor immune response and long-term benefits is still an urgent clinical issue.

Previous studies have confirmed that the Newcastle disease oncolytic virus (NDV) can selectively infect tumor cells while sparing normal cells, demonstrating an acceptable safety profile. In this study, investigators have developed a nove PIN . Preclinical studies have shown that combining PIN with anti-PD1 therapy can reverse the immunosuppressive microenvironment and transform "cold" tumors into "hot" tumors, thereby triggering local and systemic anti-tumor immune responses and significantly improving the efficacy of the immune checkpoint inhibitor(ICI). Based on these preclinical findings, investigators are conducting this clinical trial to evaluate the safety and anti tumor activity of the PIN and anti-PD1 combination therapy in vivo.

In this study, 25 to 30 subjects with refractory advanced HCC will be enrolled. The initial dose for the first cycle will be determined as 4e9 or 8e9 viral particles based on the number of injectable lesions, their longest diameter, and the tumor volume capacity.

Following the first cycle of treatment, the subsequent dose and injection sites of PIN will be adjusted based on the permissible volume of the injected tumor mass, according to the following principles:

PIN injection frequency: day 0 and day 3, per 3 weeks for 8 cycles; unless unavailability of injection lesion, disease progression (PD) or serious intolerable adverse events (AEs).

PIN injection dosage:

1. a.For patients with a single injectable lesion with a maximum diameter of <8 cm, the initial cycle's PIN dose is 4e9 viral particles. Subsequent cycles will maintain this dose of 4e9 or increase it to 8e9 viral particles based on the lesion's capacity to accommodate the injection volume; b. For patients with a single injectable lesion with a maximum diameter of ≥8 cm, the initial cycle's PIN dose is 8e9 viral particles. Subsequent cycles will maintain this dose of 8e9 viral particles based on the lesion's capacity to accommodate the injection volume.
2. a.For patients with two injectable lesions, injections will alternate between the two lesions after two cycles. The initial cycle's PIN dose is 4e9 viral particles, and the second cycle will maintain this dose of 4e9 or increase it to 8e9 viral particles based on the tumor volume's capacity; b.For patients with injectable lesions with a maximum diameter of ≥8 cm, the initial cycle's PIN dose is 8e9 viral particles, and subsequent cycles will maintain this dose of 8e9 or decrease it to 4e9 viral particles based on the lesion's capacity.
3. a.For patients with multiple injectable lesions (≥ 3), after 1-2 cycles of injections in each injectable lesion, injections are alternated between lesions. The initial injection dose for each lesion is determined by the size of the lesion; b.For lesions <3 cm, the initial cycle's dose is 4e9 viral particles, and the second cycle will maintain this dose of 4e9 or increase it to 8e9 viral particles based on the tumor volume's capacity; c.For lesions ≥3 cm, the initial cycle's injection dose is selected as 8e9 viral particles, and subsequent cycles will maintain this dose of 8e9 or decrease it to 4e9 viral particles based on the tumor volume's capacity.
4. After injections, if the tumor shrinks by 0.5-1 cm in diameter, the injection dose should be adjusted to 2e9 viral particles until the tumor disappears.

Anti-PD1 infusion frequency: day -3, per 3 weeks for 8 cycles; until unacceptable toxicity occurred or PD.

Objectives:

The primary objective are to assess the safety and adverse event profile of the combination regimen.

The coprimary objective is immune response, assessed by CD8+T cells with special phenotype by Fluorescence Activating Cell Sorter (FACS). The secondary objectives are to evaluate disease control rate (DCR), objective response rate (ORR), duration of response (DOR), progression-free survival (PFS), overall survival (OS), and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 (inclusive).
2. Eastern Cooperative Oncology Group (ECOG) performance status ≤2 and Estimated life expectancy of more than 3 months.
3. Histopathological /cytological or diagnosed clinically confirmed locally advanced or metastatic HCC having undergone treatments recommended by the "Primary Liver CancerDiagnosis and Treatment Guidelines (2024 Edition)" ,which is refractory/relapsed after and/or intolerant of standard therapies (including targeted therapy and immunotherapy) or for which no subsequent standard therapy exists.
4. At least one measurable lesion at baseline according to investigators Response Evaluation Criteria in Solid Tumours 1.1 (RECIST 1.1).
5. Patients with injectable lesions (those suitable for direct injection or injection with the assistance of medical imaging), defined as follows: at least one injectable lesion in the skin, mucous membrane, subcutaneous tissue, lymph node or visceral organ with a longest diameter ≥10 mm.
6. Subjects are willing to accept tumor rebiopsy in the process of this study.
7. Barcelona Clinic Liver Cancer (BCLC) stage ≤C.
8. Adequate organ function as defined by the following criteria:

   * Absolute neutrophil count (ANC) ≥ 1 x 10^9/L, Platelet count ≥50 x 10^9/ L, hemoglobin (Hgb) ≥ 80g/L ;
   * Serum creatinine≤1.5 upper limit of normal (ULN) or creatinine clearance (as estimated by Cockcroft Gault) ≥60 mL/min;
   * Serum aspartate amino transferase (AST) and alanine aminotransferase (ALT), ≤5 x ULN ; Total serum bilirubin ≤3 x ULN);
   * Cardiac ejection fraction ≥ 50%, no evidence of pericardial effusion as determined by an echocardiogram (ECHO), and no clinically significant electrocardiogram (ECG) findings;
   * International Normalized Ratio (INR) ≤ 1.5 times the upper limit of normal (ULN), and Activated Partial Thromboplastin Time (APTT) ≤ 1.5 times ULN;
   * Baseline oxygen saturation >91% on room air.
9. • Patients with chronic or acute hepatitis B virus (HBV) infection [ as characterized by positive hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibodies (anti-HBcAb) with detectable HBV DNA (≥20 IU/ml) ] must receive effective antiviral treatment before enrollment and during the treatment period, and their HBV DNA levels must be dynamically monitored during each treatment cycle.

   * Patients who test positive for anti-hepatitis B core (HBc) with undetectable HBV DNA (<20 IU/ml) do not require anti-viral therapy prior to enrollment.however, these subjects will be tested at every cycle to monitor HBV DNA levels and initiate antiviral therapy if HBV DNA is detected (≥20 IU/ml).
   * Subjects with chronic infection by hepatitis C virus (HCV), who are untreated, are allowed on study. In addition, subjects with successful HCV treatment are allowed, as long as 4 weeks have passed between completion of HCV therapy and start of study drug.
10. Previous treatments must be completed for more than 4 weeks prior to the enrollment of this study, and subjects have recovered to <= grade 1 Toxicity (except for hematological toxicities and clinically non-significant toxicities such as alopecia).
11. Pregnancy tests for women of childbearing age shall be negative; Both men and women agreed to use effective contraception during treatment and during the subsequent 1 year.
12. Voluntarily participate in this clinical trial and sign an informed consent form.

Exclusion Criteria:

1. Subjects are being treated with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of enrollment.
2. Active central nervous system disease involvement (but allow patients with prior brain metastases treated at least 4 weeks prior to enrollment that are clinically stable and do not require intervention), or prior history of Common Terminology Criteria for Adverse Events (CTCAE) Grade ≥3 drug-related Central Nervous System (CNS) toxicity.
3. Presence or suspicion of fungal, bacterial, viral, or other infection that is uncontrolled or requiring intravenous (IV) antimicrobials for management.
4. Any serious underlying medical (eg, pulmonary, renal, hepatic,gastrointestinal, or neurological) or psychiatric condition or any issue that would limit compliance with study requirements.
5. Major surgery or trauma occurred within 28 days prior to enrollment, or major side effects have not been recovered.
6. Received cytotoxic chemicals, monoclonal antibodies, immunotherapy or other intervene within 4 weeks or 5 half-lives before enrollment.
7. Received radiotherapy within 3 months before enrollment.
8. Patients with primary immunodeficiency or autoimmune diseases requiring immunosuppressive therapy.
9. The presence of uncontrollable serous membrane fluid, such as massive pleural effusion or ascites.
10. Previous or concurrent cancer within 3 years prior to treatment start except for curatively treated cervical cancer in situ, non-melanoma skin cancer, superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor invades lamina propria)].
11. Known positive test result for human immunodeficiency virus (HIV) or acquired immune deficiency syndrome (AIDS).
12. Prior organ allograft transplantations or allogeneic hematopoietic stem cell transplantation.
13. History of allergy or intolerance to study drug components.
14. Pregnant or breast-feeding. Women of childbearing potential must have a pregnancy test performed within 7 days before the enrollment, and a negative result must be documented.
15. Being participating any other trials or withdraw within 4 weeks.
16. Researchers believe that other reasons are not suitable for clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related AEs | Up to 12 months since the initiation of treatment.
  Treatment-related AEs are defined as any adverse medical events occurring since the initiation of treatment and grading these toxicities by Common Terminology Criteria for Adverse Events (CTCAE) V5.0.

SECONDARY OUTCOMES:
DCR | Up to 2 years since the initiation of treatment.
  DCR includes complete response (CR) ,partial response (PR) and stable disease (SD) defined by investigators according to Immune Response Evaluation Criteria in Solid Tumours (iRECIST) criteria or modified Response Evaluation Criteria in Solid Tumours (mRECIST) criteria.
ORR | Up to 2 years since the initiation of treatment.
  ORR includes CR and PR defined by investigators according to iRECIST or mRECIST criteria.
DOR | Up to 5 years since the initiation of treatment.
  DOR is defined as the date of their first CR or PR (which is subsequently confirmed) to PD assessed by investigators, or death regardless of cause.
PFS | Up to 5 years since the initiation of treatment.
  PFS is defined as the time from the initiation of treatment to the date of PD assessed by investigators, or death any cause. Participants not meeting the criteria for progression by the analysis data cutoff date were censored at their last evaluable disease assessment date.
OS | Up to 5 years since the initiation of treatment.
  OS is defined as the time from the initiation of treatment to the date of death. Subjects who have not died by the analysis data cutoff date will be censored at their last contact date.
Quality of Life Assessment. | Every 6 weeks up to 2 years since the initiation of treatment.
  Quality of life will be evaluated by European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ)-Core 30 (C30) a core scale for all cancer patients, with a total of 30 items. Among them, items 29 and 30 are divided into seven levels. Based on the responses of the subjects, they are scored from 1 to 7 points. Other items are divided into four levels: never, a little, quite a bit, and a lot. When scoring, directly assign a score from 1 to 4 points.The researchers will assess changes in quality of life by calculating total scores.

OTHER OUTCOMES:
Immunological response | PB samples are collected at least on day 0 (before PIN injection), 2, 3 (before PIN injection) and 5 during each treatment cycle ( each cycle is 21 days).
  Dynamics and molecular characteristics of CD8+ T cells with special phenotypes induced by PIN injection and its association with the treatment outcome. The relationship between the number of the CD8+ T cells and its anti-tumor effect was analyzed. To analyze the number and function of the CD8+ T cells in PB of patients with primary or acquired resistance after PIN injection and to summarize the key cellular and molecular mechanisms of resistance.
The level of cytokines and anti-PIN antibodies in serum . | PB samples are collected at least on day 0 (before PIN injection), 2, 3 (before PIN injection) and 5 during each treatment cycle ( each cycle is 21 days).
  The cytokines mainly include interleukin-1beta (IL-1β ) (pg / ml), IL-2(U/ml), IL-6(pg / ml),IL-10(pg / ml), tumor necrosis factor-α (TNF-α)(pg / ml), et al.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Han, Ph.D, Study Director — Biotherapeutic Department, Chinese PLA General Hospital; Lilin Ye, Ph.D, Study Director — Department of Tumor Immunology, Changping Laboratory; Zhijun Wang, M.D, Study Director — Department of Interventional radiology, Chinese PLA General Hospital; Guanghua Rong, Ph.D, Study Director — Biotherapeutic Department, the Fifth Medical Center of the PLA General Hospital
Locations (1):
- China, Beijing, Biotherapeutic Department of Chinsese PLA Gereral Hospital, China